CLINICAL TRIAL: NCT01297556
Title: Examining Patient Attributes To Determine Optimal Treatment Outcome in Irritable Bowel Syndrome.
Brief Title: Patient Attributes for Optimal Treatment Outcome in Irritable Bowel Syndrome.
Acronym: IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michigan Gastroenterology Institute (Other)
Responsible Party: Iftiker Ahmad, M.D., Michigan Gastroenterology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MGI-IKA-IBS-2011
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Patients in this group will receive conventional treatment for IBS, including anti-diarrhea agents, laxatives, bulking agents and anti-spasmodic.
- Treatment (Experimental): Patients in this group will receive conventional treatment for IBS, but in addition will receive 6 weeks of CBT
  Interventions: Behavioral: Cognitive Behavior Therapy(CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy(CBT) — Cognitive Behavior Therapy(CBT) for 6 weeks.
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine if any specific patient characteristics lead to improved outcome of IBS treatment, when conventional treatment as well as Cognitive Behavioral Therapy is used in combination.

DETAILED DESCRIPTION:
Although research has demonstrated the efficacy of various psychological and pharmacological treatments for irritable bowel syndrome (IBS)1, health professionals have limited information about how to determine which specific treatment regimens lead to optimal outcomes for specific IBS populations 2,3. A prevalent syndrome, with high healthcare costs, IBS is a debilitating chronic functional bowel disorder with increasingly interconnected psychosocial and gastrointestinal afflictions4. In general, IBS sufferers have not been found to respond consistently to a single medication or class of medications5. In the wake of the failures of medical therapies, many psychological interventions, adjunct to standard IBS treatments, have been examined1,6 such as Blanchard and Scharff's 2002 review of 12 random controlled trials that found strong evidence for the utility of hypnotherapy, cognitive behavioral therapy (CBT), and brief psychodynamic psychotherapy in helping to alleviate IBS symptoms7. Similarly, in a more recent study involving a meta-analysis of seventeen studies, with randomized trials comparing classes of psychological interventions, found that these psychological treatments also play a role in improving quality of life of IBS suffers1. Among these psychological interventions, cognitive behavioral therapy (CBT), a prescriptive therapy that specifically targets faulty thinking patterns, has been found to be quite effective in many empirical investigations. Recent evaluations of CBT interventions have found the therapy to have a direct effect on global improvements of IBS symptoms and quality of life8. Despite its demonstrated effectiveness, however, CBT does not work for all patients3,6,8. The successes of medical therapy alone compared to a treatment regimen combining psychological and pharmaceutical interventions have been greeted with mixed results- leading to the unnecessary waste of health resources in the course of treatment3,6. To decrease medical costs, as well to foster optimal treatment for IBS patients, there is a need for a better method of identifying which patients will most benefit from specific treatment options s (i.e. conventional medical treatment versus standard treatment and CBT)2,3.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed IBS patients using Rome III criteria above the age of 18.

Exclusion Criteria:

* Patients with non-functional GI disorders, severe psychiatric disorders, including psychotic disorders, actively suicidal or alcoholism/other drug dependencies.
* Pregnant women and minors(under age 18) will also be excluded.
* Prisoners will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
IBS Quality of Life Inventory(IBS QOLF) | 6 months
  Significant improvement in IBS QOLF score in the treatment group

SECONDARY OUTCOMES:
Behavioral Symptom Inventory | 6 months
  improvement in emotional function

CONTACTS AND LOCATIONS:
Overall Officials: Iftiker Ahmad, M.D., Principal Investigator — Michigan Gastroenterology Institute
Locations (1):
- Michigan Gastroenterology Institute, East Lansing, Michigan, United States

REFERENCES:
- [Background] 1. Lackner JM, Mesmer C, Morley S, Dowzer C, Hamilton S. Psychological Lackner JM, Mesmer C, Morley S, Dowzer C, Hamilton S. Psychological Treatments for Irritable Bowel Syndrome: A Systematic Review and Meta-Analysis. J Consult Psychol. 2004;72(6):1100-1113. 2. Spiller R, Aziz Q, Creed F, et al. Guidelines on the irritable bowel syndrome: mechanisms and practical management. Gut. 2007;56(12):1770-98. 3. Zijdenbos IL, de Wit NJ, van der Heijden GJ, Rubin G, Quartero AO. Psychological treatments for the management of irritable bowel syndrome. Cochrane Database Syst Rev. 2009;(1):CD006442. 4. Jones R, Latinovic R, Charlton J, Gulliford M. Physical and psychological co-morbidity in irritable bowel syndrome: a matched cohort study using the General Practice Research Database. Aliment Pharmachol Ther. 2006;24(5):879-886. 5.Jailwala J, Imperiale TF, Kroenke K. Pharmacologic treatment of the irritable bowel syndrome: a systematic review of randomized, controlled trials. Ann Intern Med. 2000 Jul 18;133(2):136-47. Review. PMID: 10896640 6. 6. Spanier JA, Howden CW, Jones MP. A Systematic Review of Alternative Therapies in the Irritable Bowel Syndrome. Arch Intern Med. 2003;163(3):265-674. 7.Blanchard EB, Scharf L. Psychosocial aspects of assessment and treatment of irritable bowel syndrome in adults and recurrent abdominal pain in children. J Consult Psychol. 2002;70(3):725-738. 8. Lackner JM, Jaccard J, Krasner SS, Katz LA, Gudleski GD, Blanchard EB. How does cognitive behavior therapy for irritable bowel syndrome work? A mediational analysis of a randomized clinical trial. Gastroenterology. 2007 Aug;133(2):433-44. Epub 2007 May 21. PMID: 17681164